CLINICAL TRIAL: NCT03074747
Title: The Comparison of Different Questionnaires for Preoperative Screening and Perioperative Risk Prediction in Obstructive Sleep Apnea Patients in China
Brief Title: Comparison of Four Questionnaires for OSA Screening in China
Acronym: COQ
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CT2016
Record Dates: First submitted 2017-02-22; First posted 2017-03-09 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Organic Obstructive Sleep Apnea (Diagnosis); Questionnaire; Chiari Malformation
MeSH Terms: conditions — Disease; Arnold-Chiari Malformation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: questionnaires — After filled the questionnaires, the patients will receive the PSG monitoring

SUMMARY:
Background: Obstructive sleep apnea (OSA) refers to the apnea and hypopnea caused by upper airway obstruction during sleep. Patients are associated with sleep disorders, frequent desaturation, hypertension, coronary heart disease, cerebrovascular disease and diabetes. OSA prevalence increased in China in recent years. It is estimated that nearly 80% of men and 93% of women are not diagnosed for moderate and severe OSA. Anesthesiologists and surgeons paid more attention on those high risk patients. The gold standard for OSA diagnosis is apnea and hypopnea index (AHI) obtained from polysomnography (PSG). But it is difficult to carry out PSG regularly in primary health care institutions in China for its high cost and long waiting list. So many OSA questionnaires are developed in Europe and North America, obesity is an important risk factor for OSA for them. But in China people have different anatomical characteristics, the diagnosis sensitivity and specificity of those methods has not been reported in China.

Methods and Design: Participants for this study will be recruited in Beijing Tongren Hospital scheduled for elective surgery under general anesthesia. A total of 1200 adult male patients will be enrolled. It is including 3 kinds of persons. 1. To accept PSG monitor in sleep center. 2. To receive OSA correction surgery (UPPP). 3. To receive ophthalmological surgery under general anesthesia.

Detailed inquiry and record all medical history. Upper airway assessment will be recorded. Preoperative snoring questionnaires will be integrated according to the four questionnaires. All patients complete PSG monitor. For patients undergoing surgical treatment, postoperative continuous pulse oximetry will be recorded for 24 hours. All postoperative adverse events will be recorded.

The primary endpoint:

All the patients complete the four snoring questionnaires (ASA, Berlin, STOP and STOP-BANG) before PSG test.

The secondary endpoints:

PSG monitor will be completed before operation. Medical history, upper airway assessment, postoperative 24 hours continuous pulse oximetry monitor and all perioperative adverse events will be recorded.

The purpose is to compare the specificity and sensitivity of four questionnaires to figure out OSA. To find suspected OSA patients before operation with one easy-to-use assessment questionnaire and direct OSA clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (18-60ys)
2. Male
3. ASA Ⅰ～Ⅲ grade
4. Applie to receive PSG monitor in sleep center
5. Plan to receive ophthalmological surgery under general anesthesia
6. To accept OSA correction surgery (UPPP)

Exclusion Criteria:

1. Severe maxillofacial deformities, pharyngeal reconstruction surgery history ( velopharynoplasty, upper and lower jaw orthopedic surgery, cleft lip and palate surgery)
2. Disturbance of consciousness, no self-control ability, serious mental illness, long-term alcohol abuse, drug abuse
3. Took mental or nervous system drugs within 3 months
4. Sleep apnea caused by hypothyroidism, acromegaly, laryngeal spasm, vocal cord paralysis
5. Epilepsy, neuromuscular disease
6. central sleep apnea
7. Ventilator treatment before monitor for more than 1 month
8. Llliteracy
9. Non-Chinese

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants for this study will be recruited Beijing Tongren Hospital scheduled for elective surgery under general anesthesia. A total of 1200 adult male patients will be enrolled. It is including 3 kinds of persons.
  1. To accept PSG monitor in ENT sleep center.
  2. To accept OSA correction surgery (UPPP).
  3. To receive the ophthalmological surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-03 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Berlin questionnair | From randomization to complete PSG monitor, assessed up to 3 months
  The final reports of the questionnaire
ASA Checklist | From randomization to complete PSG monitor, assessed up to 3 months
  The final reports of the questionnaire
STOP Questionnaire | From randomization to complete PSG monitor, assessed up to 3 months
  The final reports of the questionnaire
STOP-Bang Scoring Model | From randomization to complete PSG monitor, assessed up to 3 months
  The final reports of the questionnaire

SECONDARY OUTCOMES:
PSG monitor | on the day of PSG reservation or before operation
  golden standard for OSA diagnosis

OTHER OUTCOMES:
Medical history | From randomization to complete PSG monitor, assessed up to 3 months
  to learn about the medical history
upper airway assessment | From randomization to complete PSG monitor, assessed up to 3 months
  for the difficult airway evaluate and management
adverse events | during the induction of anesthesia, the whole period of anesthesia, in PACU and postoperative 24 hours
  to record the related adverse events during the perioperative period
continuous pulse oximetry monitor | postoperative 24 hours, continuous
  To monitor the saturation after surgery for the first 24 h

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stradling JR, Davies RJ. Sleep. 1: Obstructive sleep apnoea/hypopnoea syndrome: definitions, epidemiology, and natural history. Thorax. 2004 Jan;59(1):73-8. doi: 10.1136/thx.2003.007161. PMID 14694254
- [Result] Chung SA, Yuan H, Chung F. A systemic review of obstructive sleep apnea and its implications for anesthesiologists. Anesth Analg. 2008 Nov;107(5):1543-63. doi: 10.1213/ane.0b013e318187c83a. PMID 18931212
- [Result] Joshi GP, Ankichetty SP, Gan TJ, Chung F. Society for Ambulatory Anesthesia consensus statement on preoperative selection of adult patients with obstructive sleep apnea scheduled for ambulatory surgery. Anesth Analg. 2012 Nov;115(5):1060-8. doi: 10.1213/ANE.0b013e318269cfd7. Epub 2012 Aug 10. PMID 22886843
- [Result] Adesanya AO, Lee W, Greilich NB, Joshi GP. Perioperative management of obstructive sleep apnea. Chest. 2010 Dec;138(6):1489-98. doi: 10.1378/chest.10-1108. PMID 21138886
- [Result] Turner K, VanDenkerkhof E, Lam M, Mackillop W. Perioperative care of patients with obstructive sleep apnea - a survey of Canadian anesthesiologists. Can J Anaesth. 2006 Mar;53(3):299-304. doi: 10.1007/BF03022219. PMID 16527797
- [Result] Mickelson SA. Preoperative and postoperative management of obstructive sleep apnea patients. Otolaryngol Clin North Am. 2007 Aug;40(4):877-89. doi: 10.1016/j.otc.2007.04.007. PMID 17606028
- [Result] American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Practice guidelines for the perioperative management of patients with obstructive sleep apnea: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Anesthesiology. 2014 Feb;120(2):268-86. doi: 10.1097/ALN.0000000000000053. No abstract available. PMID 24346178
- [Result] Fischer MK, Martinez D, Cassol CM, Rahmeier L, Vieira LR. Immediate and overnight recumbence-dependent changes of neck circumference: relationship with OSA severity in obese and nonobese subjects. Sleep Med. 2012 Jun;13(6):650-5. doi: 10.1016/j.sleep.2012.02.007. Epub 2012 Mar 17. PMID 22425575
- [Result] Franklin KA, Lindberg E. Obstructive sleep apnea is a common disorder in the population-a review on the epidemiology of sleep apnea. J Thorac Dis. 2015 Aug;7(8):1311-22. doi: 10.3978/j.issn.2072-1439.2015.06.11. PMID 26380759
- [Result] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. Validation of the Berlin questionnaire and American Society of Anesthesiologists checklist as screening tools for obstructive sleep apnea in surgical patients. Anesthesiology. 2008 May;108(5):822-30. doi: 10.1097/ALN.0b013e31816d91b5. PMID 18431117
- [Result] Chung F, Subramanyam R, Liao P, Sasaki E, Shapiro C, Sun Y. High STOP-Bang score indicates a high probability of obstructive sleep apnoea. Br J Anaesth. 2012 May;108(5):768-75. doi: 10.1093/bja/aes022. Epub 2012 Mar 8. PMID 22401881